CLINICAL TRIAL: NCT01124474
Title: Evaluation of the Use of Arterial Pulse Waveform Contour Analysis for Goal Directed Therapy in Patients Undergoing Major Spine Surgery
Brief Title: Arterial Pulse Waveform Contour Analysis for Intraoperative Goal Directed Therapy in Major Spine Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was stopped because of lack of posterior only major spine surgeries.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5100118
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Surgical Procedures, Operative
MeSH Terms: interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard fluid management (No Intervention): Standard intraoperative fluid management as determined by usual monitoring and decision making applied by anesthesiology team
- Vigileo model number MHM1 (Other): Pulse contour waveform analysis derived stroke volume variation will be used to guide intraoperative fluid administration. Additional fluid boluses will be given to the patient when SVV>12%.
  Interventions: Other: goal directed therapy

INTERVENTIONS:
Other: goal directed therapy — Pulse contour waveform analysis derived stroke volume variation will be used to guide intraoperative fluid administration. Additional fluid boluses will be given to the patient when SVV>12%.
  Arms: Vigileo model number MHM1

SUMMARY:
This study evaluates whether using information from a special arterial blood pressure monitor to guide how much fluid is given during surgery changes how long a patient stays in the hospital after the surgery. There is scientific evidence from using similar information from different devices that this technique might allow us to do a better job giving fluids during surgery and that this may be associated with a shorter hospital stay after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for major spine surgery at LLUMC University Hospital will be eligible for participation in this study

Exclusion Criteria:

* age under 18yr,
* coagulopathy, significant renal or hepatic dysfunction (creatinine or liver enzymes > 50% above normal values),
* congestive heart failure,
* cardiac arrhythmias producing irregular rhythms, and patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Use of Arterial Pulse Waveform Contour Analysis for Goal Directed Therapy in Patients Undergoing Major Spine Surgery | From end of surgey to approximately 1 week
  time in days from the end of surgery to hospital discharge

SECONDARY OUTCOMES:
Evaluation of the Use of Arterial Pulse Waveform Contour Analysis for Goal Directed Therapy in Patients Undergoing Major Spine Surgery | from the end of surgery to approximately 1 month
  The measure of quality of recovery using scoring system; assessed by patient and nursing team

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate, M.D., Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States